CLINICAL TRIAL: NCT01540396
Title: GD2M Study:Gestational Diabetes Diagnostic Methods
Brief Title: Gestational Diabetes Diagnostic Methods
Acronym: GD2M
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: PRO11080682
Record Dates: First submitted 2012-02-15; First posted 2012-02-28 (Estimated); Last update posted 2016-02-04 (Estimated); Status verified 2016-02

CONDITIONS: Gestational Diabetes
Keywords: Gestational Diabetes
MeSH Terms: conditions — Diabetes, Gestational | interventions — Diet Therapy; Dosage Forms

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 75 Gram OGTT (Active Comparator): The 2011 ADA criteria will be used to diagnose gestational diabetes in this study arm.
  Interventions: Behavioral: Dietary modification and medications
- 100 gram OGTT (Active Comparator): A 2 step approach to the diagnosis of gestational diabetes will be used in this arm. Patients who have a 50 gram, 1 hour glucose challenge test result greater than 135 mg/dL will be diagnosed with gestational diabetes if their 3 hour, 100 gram OGTT results exceed the diagnostic threshold recommended by Carpenter and Coustan.
  Interventions: Behavioral: Dietary modification and medications

INTERVENTIONS:
Behavioral: Dietary modification and medications — Patients diagnosed with gestational diabetes will receive dietary advice and instruction on blood glucose monitoring from their regular prenatal doctors, consistent with standard of care practices. Medications (glyburide, insulin) will be used as needed to assist with blood glucose control.

SUMMARY:
This is a pilot feasibility study of 40 pregnant women to test the investigators' recruitment, enrollment and randomization procedures in preparation to conduct a larger randomized control trial to compare diagnostic methods for gestational diabetes. The two methods that are being compared are the 2 hour 75 gram OGGT (2011 ADA guidelines) versus a 1 hour 50 gram GCT + 3 hour 100 gram OGTT if the 1 hour result is abnormal (Carpenter and Coustan criteria).

DETAILED DESCRIPTION:
This is a pilot feasibility study of 40 pregnant women between 24-28 weeks gestation to test the investigators recruitment, enrollment and randomization procedures in preparation to conduct a larger randomized control trial to compare diagnostic methods for gestational diabetes.

Forty women 18 years of age or older will be recruited at 20-24 weeks pregnancy from the ob/gyn outpatient practices at Magee-Women's hospital (MWH). Eligible women will return to MWH main lab between 24-28 weeks gestation for the routine 1 hour 50gm glucose challenge test. Women with blood glucose values less than 200 will be randomized to receive either the fasting 2 hour 75 gm oral glucose tolerance test (OGTT)or the 3 hour 100 gm OGGT within two weeks. Gestational diabetes will be determined for the 2 hour 75 gm OGGT arm based on the 2011 ADA guidelines and the 3 hour 100 gm OGGT arm based on the Carpenter and Coustan criteria. Patients and their providers will be informed of the diagnosis of gestational diabetes, but they will be blinded to the criteria used to make the diagnosis as well as the specific results of glucose tolerance testing.

Chart reviews will be conducted to assess for perinatal maternal and infant health factors (e.g.pregnancy weight, gestational weight gain, co morbidities) as well as for data on perinatal outcomes related to GDM such as macrosomia, c-sections, and birth trauma. Two brief self-administered questionnaire will assess participants' views on screening for gestational diabetes and assess participants experience with and solicit feedback on the study procedures.

At the end of this pilot study, the investigators will have experience with recruitment, retention, and randomization procedures and have made the necessary protocol revisions. If successful, this feasibility study will provide the preliminary data and feasibility justification needed to conduct a larger randomized control trial to compare the effectiveness of two diagnostic methods for gestational diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Singleton pregnancy
* Plan to undergo gestational diabetes screening at 24-28 weeks' gestation.

Exclusion Criteria:

* Existing Type 1 or Type 2 diabetes
* Diabetes diagnosed early in pregnancy (less than 24 weeks gestation)
* Multiple gestation (e.g. twins, triplets)
* Chronic hypertension (requiring medications)
* Oral, IM or IV corticosteroid use within the previous 30 days
* Major congenital anomaly or anticipated preterm delivery before 28 weeks
* Inability to complete 50 gram GCT before 28 completed weeks' gestation
* Patients with known HIV, Hepatitis B or C virus.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 47 (Actual)
Dates: Start 2012-02; Primary Completion 2013-02 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Macrosomia | Will be assessed from study enrollment until delivery (approximtaly 40 weeks' gestation)
  Defined as birthweight >90th percentile for gestational age or birthweight >4000 grams
Cesarean delivery | Will be assessed from study enrollment until delivery (approximtaly 40 weeks' gestation)
  Primary or repeat cesarean delivery
Diagnosis of gestational diabetes | Will be followed from study enrollment until delivery (approximately 40 weeks' gestation)
  Assess how frequently a diagnosis of gestational diabetes is made

SECONDARY OUTCOMES:
Pre-eclampsia or gestational hypertension | Will be assessed from study enrollment until 30 days after delivery
  New onset hypertension +/- proteinuria
Neonatal hypoglycemia | First 24 hours of life
  Defined as blood glucose less than 80 mg/dL from heel stick within 1 hour after delivery
Neonatal hyperbilirubinemia | First 7 days of life
  Defined as bilirubin greater than 5 mg/dL over 24 hours from heel stick
Infant birth trauma | Will be assessed from study enrollment until delivery (approximtaly 40 weeks' gestation)
  Defined as shoulder dystocia/brachial plexus injuries
Maternal birth trauma | Will be assessed from study enrollment until delivery (approximtaly 40 weeks' gestation)
  3rd or 4th degree perineal laceration or postpartum hemorrhage

CONTACTS AND LOCATIONS:
Overall Officials: Christina M Scifres, MD, Principal Investigator — University of Pittsburgh; Esa Davis, MD MPH, Principal Investigator — University of Pittsburgh
Locations (1):
- Magee-Womens Hospital, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No